CLINICAL TRIAL: NCT00412477
Title: RV 151: A Phase I Study of Safety and Immunogenicity of the WRAIR HIV-1 Vaccine LFn-p24 Administered by the Intramuscular (IM) Route in Healthy Adults, WRAIR #984, HSRRB Log # A-11905.
Brief Title: A Phase I Study of Safety and Immunogenicity of the WRAIR HIV-1 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: WRAIR 984; HSRRB Log # A-11905 (Other: USAMRMC)
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: HIV Infections
Keywords: HIV; Lfn-p24; Anthrax; IM; HIV-1; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Anthrax

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 - LFn-p24 ISOug with Alhydrogel (Experimental): HIV LFn-p24 is a combination of an Anthrax derived polypeptide Lethal factor (LFn), from which the toxin domain has been removed, and the HIV-1 gag p24 protein has been fused to LFn. Lfn-p24 is formulated in liquid form, and vialed. Product is administered IM, 1ml. Six subjects (4 vaccines and 2 placebos).
  Placebo recipients will receive a saline preparation in similar volume given IM.
  Immunizations given at 0, 4 and 16 weeks
  Interventions: Biological: HIV LFn-p24
- Group 2 - LFn-p24 300ug with Alhydrogel (Experimental): HIV LFn-p24 is a combination of an Anthrax derived polypeptide Lethal factor (LFn), from which the toxin domain has been removed, and the HIV-1 gag p24 protein has been fused to LFn. Lfn-p24 is formulated in liquid form, and vialed. Product is administered IM, 1ml. Six subjects (4 vaccines and 2 placebos).
  Placebo recipients will receive a saline preparation in similar volume given IM.
  Immunizations given at 0, 4 and 16 weeks
  Interventions: Biological: HIV LFn-p24
- Group 3 - LFn-p24 450ug with Alhydrogel (Experimental): HIV LFn-p24 is a combination of an Anthrax derived polypeptide Lethal factor (LFn), from which the toxin domain has been removed, and the HIV-1 gag p24 protein has been fused to LFn. Lfn-p24 is formulated in liquid form, and vialed. Product is administered IM, 1ml. Six subjects (4 vaccines and 2 placebos).
  Placebo recipients will receive a saline preparation in similar volume given IM.
  Immunizations given at 0, 4 and 16 weeks
  Interventions: Biological: HIV LFn-p24

INTERVENTIONS:
Biological: HIV LFn-p24 — HIV LFn-p24 is a combination of an Anthrax derived polypeptide Lethal factor (LFn), from which the toxin domain has been removed, and the HIV-1 gag p24 protein has been fused to LFn. Lfn-p24 is formulated in liquid form, and vialed at 200 µg/ml and 600 µglml. The product will be administered IM in doses ranging from 150µg to 450µg with Alhydrogel.

SUMMARY:
To evaluate the safety of LFn-p24 administered at three different doses with Alhydrogel given intramuscularly

To evaluate immune responses to LFn-p24 with Alhydrogel at three different doses given intramuscularly

DETAILED DESCRIPTION:
The study seeks to enroll healthy, vaccine naïve volunteers, 18 through 45 years old. Recruitment consists of using flyers, newspaper advertising, radio, and direct mailing at local military installations, targeting the general population of the greater Washington D.C. area.

The study's primary objective is the safety and tolerability of Lfn-p24 given IM.

Volunteers will be screened (visit 1) and enrolled within 2 to 12 weeks prior to the first vaccination. Study volunteers will receive a briefing from the Principal Investigator (PI) or a sub investigator. The briefing is followed by an opportunity for questions from the volunteers. The PI or designee will then review the consent form with potential volunteers (visit 1) and answer any questions. After review, an Informed Consent will be signed and a "Test of Understanding" will be completed by all volunteers, prior to enrollment in the study. A second pre-screening visit (visit 2) will occur 3 - 30 days prior to the first vaccination (visit 3) to confirm eligibility for vaccination. During this visit each volunteer will have an opportunity to ask questions about the study.

On the day of vaccination (visits 3, 6, and 10), volunteers will be observed for 30 minutes following injection for acute adverse experiences and will be contacted the day following injection for a brief adverse reaction interview. In addition, volunteers will complete diaries for 7 days following each vaccination and will be evaluated by a clinical investigator if significant symptoms are reported. Adverse effects and laboratory abnormalities will be tabulated. Routine measurements of hematology, serum chemistry, and urinalysis laboratory tests will be performed in subsequent safety and general follow up visits.renee

LFn-p24 with Alhydrogel adjuvant will be delivered IM in the deltoid muscle at the intervals shown below. Groups will be enrolled in staggered fashion beginning with the lowest dose group. The subsequent groups receiving higher doses will then be enrolled by the investigator if the second injection of the immediate lower dose is shown to be safe and well tolerated (< grade II toxicity), after the 2 week post vaccination follow-up visit.

IMMUNIZATION SCHEDULE

Group I Subjects *6 0:150µg LFn-p24 Alhydrogel;4th Week:150µg LFn-p24 Alhydrogel; 16th Week:150µg LFn-p24 Alhydrogel; Group II Subjects *6 0:300µg LFn-p24 Alhydrogel; 4th Week: 300µg LFn-p24 Alhydrogel; 16th Week: 300µg LFn-p24 Alhydrogel; Group III Subjects *6 0: 450µg LFn-p24 Alhydrogel; 4th Week: 450µg LFn-p24 Alhydrogel; 16th Week: 450µg LFn-p24 Alhydrogel

*Six subjects per group includes 4 vaccines and 2 placebos.

ELIGIBILITY:
Inclusion Criteria:

* Citizens of the U.S.A. who are not at high-risk for HIV infection.
* Age: 18 through 45 years of age.
* For women, negative serum pregnancy test will be required within two days prior to any injection, as well as verbal assurance that adequate contraceptive measures are applied.
* Good health as determined by medical history, physical examination, and clinical judgment.

Clinical laboratory values at screening within the following ranges:

* Hematocrit: Women: > 34%: Men >38% (Mild anemia in any potential trial volunteer who is otherwise healthy attributable by appropriate laboratory studies to thalassemia minor will not be cause for exclusion)
* White blood cell count: 3,000 to 12,000 cells/mm3
* Platelets: 125,000 to 550,000 per mm3
* Chemistry Panel: Expanded chemistry panel within institutional normal ranges or accompanied by site physician approval.
* Urine dipstick for protein and blood: negative or trace. If either is ≥ 1+, obtain complete urinalysis (UA). If microscopic UA confirms evidence of hematuria or proteinuria ≥ 1+, the volunteer is ineligible unless menstruating, then a repeat UA is required.
* Negative serology for HIV infection (ELISA test).
* Availability for at least 52 weeks
* Successful completion of the Test of Understanding, Commitment for Trial Participation and signature of the approved Trial Consent Form.

Exclusion Criteria:

* Acknowledge engaging in highest-risk behavior within 48 weeks of study entry: (i.e., active injecting drug use or having sexual intercourse with a known HIV-1 infected partner).
* Have active tuberculosis or other systemic infectious process by review of systems and physical examination.
* Have a history of immunodeficiency, chronic illness requiring continuous or frequent medical intervention, autoimmune disease, or use of immunosuppressive medications.
* Have evidence of psychiatric, medical and/or substance abuse problems during the past 48 weeks that the investigator believes would adversely affect the volunteer's ability to participate in the trial.
* Have occupational or other responsibilities that would prevent completion of participation in the study.
* Have received any live, attenuated vaccine within 60 days of study entry.
* NOTE: Medically indicated subunit or killed vaccines (e.g., Hepatitis A or Hepatitis B) are not exclusionary but should be given at least 2 weeks before or after HIV immunization to avoid potential confusion of adverse reactions.
* Acute or chronic Hepatitis caused by viral or other etiology.
* Have used experimental therapeutic agents within 30 days of study entry.
* Have received blood products or immunoglobulins in the past 12 weeks.
* Have a history of anaphylaxis or other serious adverse reactions to vaccines.
* Have previously received an HIV and/or anthrax vaccine.
* Currently enrolled in other vaccine trials.
* Are pregnant or lactating.
* NOTE: Women of child-bearing potential must be using effective contraception from the date of enrollment into the protocol.
* Have an immediate type hypersensitivity reaction to aminoglyocides, e.g., kanamycin (used to prepare the LFn-p24 vaccine).
* Are study site employees who are involved in the protocol and may have direct access to the immunogenicity results.
* Are receiving ongoing therapy with immunosuppressive therapy such as systemic corticosteroids or cancer chemotherapy.
* Are active duty military or reserves.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2004-08-20 (Actual); Primary Completion 2006-03-13 (Actual); Study Completion 2006-11-01 (Actual)

PRIMARY OUTCOMES:
Humoral: Responders to ELISA and Western Blot antibodies to HIV-1 subtype B gag p24 | Days 0, 14, 42, 70, 126, 182, 252 and 364
  An HIV-I enzyme linked immunosorbent assay (ELISA) assay will be performed as designated throughout the course of the protocol during Visits 1 through 15. If the ELISA is reactive it will be repeated and an FDA- approved HIV Western blot will be performed. If the Western blot is positive, HIV molecular diagnostics (Roche Amplicor) will be performed
Cellular: Cytotoxic T-lymphocyte (CTL) responses against subtype B gag antigen target expressed in Epstein Barr Virus (EBV) transformed autologous B cell lines. | Days 3, 14, 42, 70, 126, 182, 252, and 364
  Cytotoxic T-lymphocyte (CTL) responses against subtype B gag antigen target expressed in Epstein Barr Virus (EBV) transformed autologous B cell lines. Bulk CTL is currently defined to be positive if the HIV-1 antigen expressing targets relative to control have a specific lysis 10%. CD8+ CTL occurs when lytic activity decreases by 50% after removal of CD8 cells, while removal of CD4 cells maintains specific lysis at 5%. An analogous rule is applied for CD4+ CTL
IFN-y ELISPOT assay against HIV-gag antigen. | Days 3, 14, 42, 70, 126, 182, 252, and 364
  IFN-y ELISPOT assay using a panel of B clade gag peptides. A positive responder will be defined in accordance with other HIV Vaccine Trial Network (HVTN) definitions. For example a positive response may be defined by a significant difference between the number of IFN-g spot forming cell s (SFC)/million peripheral blood mononuclear cells (PBMC) in the presence of HIV gag antigen and no antigen. Other arbitrary definitions may be used.
IFN- ICS assay against HIV-gag antigen. | Days 3, 14, 42, 70, 126, 182, 252, and 364
  For the IFN-gamma intracellular cytokine staining (ICS) assay we will use a panel of B clade gag peptides or other appropriate gag antigens. A positive responder will be defined in accordance with the HIV Vaccine Trial Network (HVTN) definitions or other definitions as appropriate. For example a positive response may be defined as a two-fold difference between the percentage of CD3+CD8+IFN-y+ or CD3+CD4+IFN-y+ T cells in the presence of HIV gag antigen compared with no antigen
Lymphocyte proliferative responses to HIV-1 subtype B gag | Days 3, 14, 42, 70, 126, 182, 252, and 364
  Lymphocyte proliferative responses to HIV- I subtype B gag p24. The data are expressed as a Lymphocyte Stimulation Index (LSI)= (PBMC cpm + antigen/ mitogen) I (PBMC cpm+ medium)] to define antigen specificity. Individuals are arbitrarily designated as responders non-responders if their LSI is greater than or equal to 5.

SECONDARY OUTCOMES:
Humoral- Binding antibodies to LFn | Days 3, 14, 42, 70, 126, 182, 252, and 364
  Expression profile surveillance of 8000 fully annotated genes in peripheral blood mononuclear cells using the Affymetrix Human Focus GeneChip to assess sentinel genes and associated cellular processes that might be correlated with protection by the vaccine.
Neutralizing antibodies to LFn | Days 3, 14, 42, 70, 126, 182, 252, and 364
  Expression profile surveillance of 8000 fully annotated genes in peripheral blood mononuclear cells using the Affymetrix Human Focus GeneChip to assess sentinel genes and associated cellular processes that might be correlated with protection by the vaccine.
Cellular: Lymphoproliferation to LFn | Days 3, 14, 42, 70, 126, 182, 252, and 364
  Expression profile surveillance of 8000 fully annotated genes in peripheral blood mononuclear cells using the Affymetrix Human Focus GeneChip to assess sentinel genes and associated cellular processes that might be correlated with protection by the vaccine.

OTHER OUTCOMES:
and Systemic Reactions After Immunization of of Lfn-p24 Given IM | 30 minutes and 7 days post vaccination
  Safety and tolerability of Lfn-p24 given IM. Adverse effects will be tabulated. Subjects will be observed for 30 minutes following immunization for evidence of immediate local and systemic reactions. They will be instructed to maintain a diary for local and systemic reactions for 7 days post-immunization and will be evaluated by a clinical investigator if significant symptoms are reported.

CONTACTS AND LOCATIONS:
Overall Officials: CDR Shirley Lee-Lecher, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Vaccine Clinical Research Center, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. UNAIDS/WHO. Report on the global HIV/AIDS epidemic.June 2000. 2. Quinn TC. Global burden of the HIV pandemic. Lancet.1996;348:99-106. 3. Moss B. Genetically engineered poxviruses for recombinant gene expression, vaccination, and safety. PNAS 1996;93; 11341-8. 4. Tartaglia J, Excler JL, El Habib R, Limbach K, Meignier B, Plotkin S, Klein M. Canarypoxvirus-based vaccines : prime-boost strategies to induce cell-mediated and humoral immunity against HIV. AIDS Res Hum Retroviruses 1998;14(supp.3): S291-S298. 5. Girard M, Excler JL. Human Immunodeficiency virus. In Vaccines. Plotkin SA and Mortimer EA Eds. Saunders, Philadelphia,1999, pp.928-967. 6. Excler J-L, Plotkin S. The prime-boost concept applied to HIV preventive vaccines. AIDS 1997;11(suppl A):S127-137. 7. Ogg GS, Jin X, Bonhoeffer S, Dunbar PR, Nowak MA, Mopnard S, Segal JP, Cao Y, 8. Rowland-Jones SL, Cerundolo V, Hurley A, Markowwitz M, Ho DD, Nixon DF, McMichael AJ. Quantitation of HIV-1-specific cytotoxic T lymphocytes and plasma load of viral RNA. Science 1998; 279: 2103-6. 8. Schmitz JE, Kuroda MJ, Santra S, Sasseville VG, Simon MA, Lifton MA, Racz P, Tenner-Racz K, Dalesandro M, Scallon BJ, Ghrayeb J, Forman MA, Montefiori DC, Rieber EP, Letvin NL, Reimann KA. Control of viremia in simian immunodeficiency virus infection by CD8 lymphocytes. Science 1999; 283: 857-60. 9. Brodie SJ, Lewinsohn DA, Patterson BK, Jiyamapa D, Krieger J, Corey L, Greenberg P, Riddell SR. In vivo migration and function of transferred HIV-1-specific cytotoxic T cells. Nature Medicine 1999; 5: 34-41. 10. Letvin NL. Progress in development of an AIDS vaccine. Science 1998; 280: 1875-9.